CLINICAL TRIAL: NCT03817359
Title: Use of a Remifentanil-propofol Mixture in Patients With Breast Cancer Undergoing Breast Cancer Surgery: a Prospective Pilot Study
Brief Title: Use of a Remifentanil-propofol Mixture in Patients Undergoing Breast Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Meng-Fu Lai, Resident physician, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2-107-05-079
Record Dates: First submitted 2019-01-19; First posted 2019-01-25 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Anesthetics; Remifentanil; Propofol
Keywords: propofol; remifentanil; total intravenous anesthesia; breast surgery

STUDY DESIGN:
Intervention Model Description: 84 patients scheduled for breast cancer surgery were randomly allocated to receive TIVA with propofol and remifentanil separately by two TCI pump (Separate group) or with remifentanil-propofol mixture by single TCI pump (Mix group), all TCI concentration adjustments during operation were based on BIS and ANI monitor.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mix infusion using single TCI pump (Experimental): participants receive total intravenous anesthesia with remifentanil-propofol mixture by single TCI pump infusion
  Interventions: Combination Product: Remifentanil-propofol mixture
- Separate infusion using two TCI pumps (No Intervention): participants receive total intravenous anesthesia with remifentanil and propofol separately by two TCI pumps infusion

INTERVENTIONS:
Combination Product: Remifentanil-propofol mixture — Participants receive total intravenous anesthesia with remifentanil-propofol mixture by single TCI pump in intervention group. All TCI target concentration adjustments or extra bolus of propofol or remifentanil during operation were based on BIS and ANI monitor.
  Arms: Mix infusion using single TCI pump

SUMMARY:
Co-administration of propofol and remifentanil is considered to be an ideal total intravenous anesthesia technique, which is widely used in induction and maintenance of general anesthesia. Remifentanil and propofol can be mixed in polypropylene syringes for one hour with a remaining concentration of 91% in small concentrations of remifentanil. However, delivery of remifentanil-propofol mixture by target-controlled infusion(TCI) for general anesthesia in surgical procedure has not been described. Breast cancer surgery ( including modified radical mastectomy and breast-conserving surgery) is a less time-consuming procedure for patients with breast cancer with one-hour duration in our hospital. This pilot study was to examine the merit of remifentanil-propofol mixture as a GA regimen for breast cancer surgery.

DETAILED DESCRIPTION:
Previous studies has described the feasibility and safety of remifentanil-propofol mixture use in sedation of pediatric patients undergoing magnetic resonance imaging or flexible fiberoptic bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* ASA II or III
* age more than 18 years
* scheduled for breast cancer surgery under general anesthesia.

Exclusion Criteria:

* previously allergic to propofol or remifentanil
* combining other surgical procedure leading to extended operative time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2018-12-27 (Actual); Study Completion 2018-12-27 (Actual)

PRIMARY OUTCOMES:
Frequency of TCI device adjustments | during procedure
  Total times of TCI pump adjustment

SECONDARY OUTCOMES:
Mean blood pressure | at 5 minute intervals perioperatively throughout the procedure in an average of 60 minutes
  measured by non-invasive blood pressure cuff
Heart rate | at 5 minute intervals perioperatively throughout the procedure in an average of 60 minutes
  recorded by ECG and pulse oximetry
Patient satisfaction | the 1 day after operation
  Rating of satisfaction by questionnaire
postoperative analgesia rescue | An average of 30 minutes after arriving at PACU
  Analgesics use during PACU stay
Total dose of remifentanil | At the end of surgery
  total consumption of remifentanil during procedure
Total dose of propofol | At the end of surgery
  total consumption of propofol during procedure

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Fu Wu, M.D., Principal Investigator — Department of Anesthesiology, Tri-Service General Hospital
Locations (1):
- Tri-Service General hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bedocs P, Evers DL, Buckenmaier CC 3rd. Predosing Chemical Stability of Admixtures of Propofol, Ketamine, Fentanyl, and Remifentanil. Anesth Analg. 2019 Jul;129(1):e13-e15. doi: 10.1213/ANE.0000000000003772. PMID 30286006
- [Result] Berkenbosch JW, Graff GR, Stark JM, Ner Z, Tobias JD. Use of a remifentanil-propofol mixture for pediatric flexible fiberoptic bronchoscopy sedation. Paediatr Anaesth. 2004 Nov;14(11):941-6. doi: 10.1111/j.1460-9592.2004.01355.x. PMID 15500495
- [Result] Stewart JT, Warren FW, Maddox FC, Viswanathan K, Fox JL. The stability of remifentanil hydrochloride and propofol mixtures in polypropylene syringes and polyvinylchloride bags at 22 degrees-24 degrees C. Anesth Analg. 2000 Jun;90(6):1450-1. doi: 10.1097/00000539-200006000-00037. PMID 10825339